CLINICAL TRIAL: NCT03591016
Title: Prospective Observational Study of Difficult Intravenous Access in the Operating Room
Status: Completed | Type: Observational
Sponsor: Ralph Beltran (Other)
Responsible Party: Sponsor-Investigator, Ralph Beltran, Staff Anesthesiologist, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB18-00495
Record Dates: First submitted 2018-06-20; First posted 2018-07-18 (Actual); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Difficult Intravenous Access

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Difficult intravenous access: Recording number of IV attempts in the operating room prior to surgery start.
  Interventions: Other: Recording number of IV attempts

INTERVENTIONS:
Other: Recording number of IV attempts — Recording number of IV attempts in the operating room

SUMMARY:
This is an observational study only, where number of attempts to establish peripheral IV catheter placement will be recorded during procedures in all anesthetizing location on the main campus of Nationwide Children's Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients 0-18 years of age
* Having surgery at Nationwide Children's Hospital

Exclusion Criteria:

* Pre-existing IV upon arrival to the operating room

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Male and female 0-18 years old undergoing surgery with anesthesia requiring an IV.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Time it takes to insert an IV | between 1 to 30 minutes

SECONDARY OUTCOMES:
Anticipated difficulty | Baseline
  Provider's prediction of how difficult it will be to start the IV on a Likert scale of 1-10, with 10 being the most difficult.
Actual difficulty | between 1 to 30 minutes
  Provider's assessment of how difficult the actual IV insertion was on the same Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Beltran, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States